CLINICAL TRIAL: NCT02659878
Title: Incidence, Influencing Factors and Outcome of Takotsubo Cardiomyopathy in Patients Suffering From Acute Non-traumatic Subarachnoid Hemorrhage
Brief Title: Takotsubo Cardiomyopathy in Patients Suffering From Acute Non-traumatic Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, assistant lecturer anesthesiologist and intensive care specialist, University of Debrecen
Other Study IDs: HBR/052/00436-2/2015; DE RKEB/IKEB:4317-2015 (Registry Identifier: REGIONAL AND INSTITUTIONAL ETHICS COMMITTEE, CLINICAL CENTER, UNIVERSITY OF DEBRECEN)
Record Dates: First submitted 2016-01-11; First posted 2016-01-21 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Takotsubo Cardiomyopathy; Subarachnoid Hemorrhage
Keywords: Takotsubo cardiomyopathy;NT-proBNP;urine metanephrine
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: bleeding, intraventricular and/ or intracerebral hemorrhage. — Patient's age, sex, comorbidities, medications, the exact time point of bleeding, the circumstances of bleeding neurological and cardiological status are recorded, laboratory tests, Transcranial Color Doppler (TCCD), echocardiography and chest X-ray examinations are carried out within 24 hours after the patient is being admitted to the ICU.

SUMMARY:
Pupose:

Takotsubo cardiomyopathy is a rare and not well-known complication of the subarachnoid hemorrhage.

This form of heart failure, called as "broke heart" or "apical ballooning syndrome", was first described by Japanese authors at the beginning of 1990's.

1.5-2.2% of acute coronary syndrome is Takotsubo cardiomyopathy. Its predisposing factors, hypothetical parthenogenesis, diagnostic criteria and therapeutic methods are already known from the literature.

The study intends to include all patients over 18 years of age who were admitted to our clinic within 48 hours after the bleeding regardless of gender, neurological status or age.

Data to be registered within 24 hours after admittance:

Instruments:

* Intracranial blood flow characteristics:TCCD - using Transcranial Color Doppler; systolic, diastolic and mean blood flow velocity, Systolic / Diastolic ratio, pulsatility index
* ECG abnormalities: Corrected QT Interval (QTc), T wave, ST segment, arrhythmia
* Echocardiography (Ejection fraction%, exact location and degree of cardiac wall motion abnormalities) - documented with video recording

Hypothesis:

The risk of Takotsubo cardiomyopathy (TS) is increased if SAH is associated with more severe state, a greater degree of bleeding, intraventricular and/ or intracerebral hemorrhage.

The definitive care of patients is postponed due to the appearance of TS, which could affect the final outcome.

DETAILED DESCRIPTION:
Data to be registered within 24 hours after admittance:

* Age of the patient
* Gender
* Comorbidities
* Currently taken medications
* The exact time point of bleeding
* Additional circumstances of the bleeding
* Physical stress factors
* Psychological stress factors
* Significant blood pressure elevation, and its assumed reason
* Severity of bleeding:Fisher's Grade; Neurological status; Hunt-Hess scale;GCS (Glasgow Coma Scale)
* Intracranial blood flow characteristics:TCCD - using Transcranial Color Doppler; systolic, diastolic and mean blood flow velocity, Systolic / Diastolic ratio, pulsatility index
* Cardiac status:Chest pain, Shortness of breath, Pulmonary edema
* ECG abnormalities: Corrected QT Interval (QTc), T wave, ST segment, arrhythmia
* Enzyme level associated with myocardial tissue necrosis: Cardiac troponin I (cTnI), creatine kinase (CK), CK-MB, Brain natriuretic peptide (BNP), N-terminal prohormone of brain natriuretic peptide (NT-proBNP)
* The amount of urine collected in 24 hours and determination of urine metanephrine, normetanephrine levels
* Chest X-ray
* Echocardiography (Ejection fraction%, exact location and degree of cardiac wall motion abnormalities) - documented with video recording
* Medication: Nimodipine, simvastatin, keeping Mg levels in the normal range, ulcer prophylaxis, painkillers
* Fluid therapy: ensuring normovolaemia

Data to be recorded during hospital stay:

* Localization of the bleeding (is there an aneurysm present, if yes what is its location, size)
* Is ventricular drain necessary?
* Treatment methods of the aneurysm:Endovascular, aneurysm clipping
* Time passed between bleeding and treatment (in hours)

The following investigations are repeated daily:

* 12-lead ECG
* Myocardial necrotic enzymes (checked daily over 1 week even if no ECG abnormalities are present) : cardiac troponin I (cTnI), creatine kinase (CK), CK-MB, Brain natriuretic peptide (BNP), N-terminal prohormone of brain natriuretic peptide (NT-proBNP)
* In case of ECG abnormalities echocardiography should take place on the same day (with video recording)
* If there are no ECG abnormalities echocardiography should be controlled once within the first week (with video recording)
* Transcranial Color Doppler (TCCD)
* Glasgow Coma Scale (GCS)
* Recording the currently used medicines with accurate doses (with special attention to the positive inotropic agents and drugs with vasoconstrictor properties)
* In case of mechanical ventilation:Fraction of inspired oxygen (FiO 2), Positive end expiratory pressure (PEEP), Blood gas analysis (PaO 2, PaCO 2), Peak pressure (PPeak)
* Noting the presence of pulmonary edema (auscultation, blood gas analysis) If Takotsubo cardiomyopathy is diagnosed, the 24-hour urine collection test should be repeated (measure the quantity of collected urine, determine urine metanephrine and normetanephrine levels)

The following diagnostic steps should be repeated after 1 month:

* Echocardiography
* 12-lead ECG
* New York Heart Association scores (NYHA scores)
* Glasgow outcome scale (GOS) - survival index
* Bartel Index, Karnofsky score - index of life quality
* The amount of urine collected in 24 hours and determination of urine metanephrine, normetanephrine levels

If echocardiography shows cardiac wall motion abnormality, cardiac examination should be carried out as the following:

* Cardiac stress test if necessary
* CT coronary angiogram if necessary
* Coronary angiography if necessary

The following examinations should be carried out after 6 months:

* Echocardiography
* 12-lead ECG
* New York Heart Association scores (NYHA scores)
* Glasgow outcome scale (GOS) - survival index
* Bartel Index
* The amount of urine collected in 24 hours and determination of urine metanephrine, normetanephrine levels

Comments:

The level of metanephrine and normetanephrine from 24-hour collected urine should be measured again after 1 and 6 months in case of patients where TS was diagnosed.

The urine of patients who have no diagnosed TS will be solely collected and serve as a control. Only 15 of these urine samples will be randomly measured to metanephrine / normetanephrine.

Patient's age, sex, comorbidities, medications, the exact time point of bleeding, the circumstances of bleeding neurological and cardiological status are recorded, laboratory tests, Transcranial Color Doppler (TCCD), echocardiography and chest X-ray examinations are carried out within 24 hours after the patient is being admitted to the ICU.

The medication to prevent vasospasm (Nimodipine, Simvastatin, sustained physiological Mg level) and ulcers, just like the drugs to relief pain are the same in case of all patients.

The goal of fluid therapy is to maintain normovolaemia. The location of the bleeding is recorded (is there any aneurysm, its size is measured; if ventricular drainage is necessary, the method that used to treat aneurysm: endovascular, clipping; time elapsed between bleeding and therapy) 12-lead ECG, cardiac enzymes, TCCD measurement, neurological state, medications and its doses, blood gas analysis in case of mechanical ventilation and ventilation parameters are carried out and recorded on a daily basis.

Cardiac ultrasound and 12-lead ECG examinations are carried out, NYHA scores, clinical outcome (GOS), quality of life (Bartel Index) and Karnofsky scores are recorded after 1 month.

If echocardiography shows cardiac wall motion abnormality, cardiac examination should be carried out as following: cardiac stress test, coronary CT angiogram and coronary angiography if necessary.

Echocardiography, 12-lead ECG examinations are repeated and NYHA scores, clinical outcome (GOS), quality of life (Bartel Index) and Karnofsky scores are recorded after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Acute subarachnoid hemorrhage
* Admittance to the neurosurgery intensive care unit within 48 hours after the bleeding has occurred
* Over 18 years of age
* No prior cardiological diseases in medical history

Exclusion Criteria:

* Known myocardial diseases (previous myocardial infarction)
* Preexisting heart failure
* Previously known structural heart disease (severe, clinically significantvalve insufficiency, and / or significant stenosis)
* Preexisting myocarditis
* Preexisting phaecromocytoma
* Preexisting hypertrophic cardiomyopathy (Left ventricle > 15 mm)
* Preexisting coronary artery stenosis that requires dilation (patients should be excluded if coronary artery stenosis with dilation need is confirmed during the follow-up period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study intends to include all patients over 18 years of age who were admitted to our clinic within 48 hours after the bleeding regardless of gender, neurological status or age.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
ECG abnormalities:Corrected QT Interval (QTc), T wave, ST segment, arrhythmia | Data to be registered within 24 hours after admittance
  12-lead ECD
ECG abnormalities:Corrected QT Interval (QTc), T wave, ST segment, arrhythmia | The following diagnostic steps should be repeated after 1 month
  12-lead ECD
urine metanephrine, normetanephrine levels | The amount of urine collected in 24 hours
  The amount of urine collected in 24 hours and determination of urine metanephrine, normetanephrine levels
urine metanephrine, normetanephrine levels | The following diagnostic steps should be repeated after 1 month
  The level of metanephrine and normetanephrine from 24-hour collected urine should be measured again after 1 and 6 months in case of patients where TS was diagnosed.
Enzyme level associated with myocardial tissue necrosis | Data to be registered within 24 hours after admittance
  Cardiac troponin I (cTnI), creatine kinase (CK), CK-MB, Brain natriuretic peptide (BNP), N-terminal prohormone of brain natriuretic peptide (NT-proBNP)
Enzyme level associated with myocardial tissue necrosis | The following diagnostic steps should be repeated after 1 month
  Cardiac troponin I (cTnI), creatine kinase (CK), CK-MB, Brain natriuretic peptide (BNP), N-terminal prohormone of brain natriuretic peptide (NT-proBNP)
Ejection fraction%, exact location and degree of cardiac wall motion abnormalities | Data to be registered within 24 hours after admittance
  Echocardiography documented with video recording
Ejection fraction%, exact location and degree of cardiac wall motion abnormalities | The following diagnostic steps should be repeated after 1 month
  Echocardiography documented with video recording

SECONDARY OUTCOMES:
New York Heart Association scores (NYHA scores) Glasgow outcome scale (GOS) - survival index Neurological status | The following examinations should be carried out after 6 months:
  Clinical outcome (GOS), quality of life (Bartel Index) and Karnofsky scores

CONTACTS AND LOCATIONS:
Overall Officials: Csilla Molnár, MD,PhD, Principal Investigator — UNIVERSITY OF DEBRECEN FACULTY OF MEDICINE Department of Anesthesiology and Intensive Care Debrecen, Hungary, 4032
Locations (1):
- UNIVERSITY OF DEBRECEN FACULTY OF MEDICINE Department of Anesthesiology and Intensive Care, Debrecen, Hajdú-Bihar, Hungary

REFERENCES:
- [Background] Castillo Rivera AM, Ruiz-Bailen M, Rucabado Aguilar L. Takotsubo cardiomyopathy--a clinical review. Med Sci Monit. 2011 Jun;17(6):RA135-47. doi: 10.12659/msm.881800. PMID 21629203
- [Derived] Molnar C, Gal J, Szanto D, Fulop L, Szegedi A, Siro P, Nagy EV, Lengyel S, Kappelmayer J, Fulesdi B. Takotsubo cardiomyopathy in patients suffering from acute non-traumatic subarachnoid hemorrhage-A single center follow-up study. PLoS One. 2022 May 26;17(5):e0268525. doi: 10.1371/journal.pone.0268525. eCollection 2022. PMID 35617162
- See also: Usefulness of MRI in takotsubo cardiomyopathy: a review of the literature Andres Alejandro Kohan1 — http://www.thecdt.org/article/view/3459/4520